CLINICAL TRIAL: NCT01116466
Title: Clinical Study to Evaluate the Implantation of the ActiGait Drop Foot Stimulator System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otto Bock Healthcare Products GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PB-SA844-100
Record Dates: First submitted 2010-04-23; First posted 2010-05-05 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-06

CONDITIONS: Stroke; Hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ActiGait (Experimental): Receiving ActiGait - implantable drop foot stimulator
  Interventions: Device: ActiGait

INTERVENTIONS:
Device: ActiGait — ActiGait - implantable drop foot stimulator

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of surgical procedure involving ActiGait - implantable drop foot stimulator.

DETAILED DESCRIPTION:
Stroke is the third leading cause of death in the United States and other developed countries and a major source of disability. Prognosis for regaining the ability to walk is good, with 64% of those initially dependent in walking regaining independence by 3 months. However, many gait abnormalities persist. A conservative estimate suggests that 20% of stroke survivors have a drop foot. Drop foot following stroke is caused by paresis of the ankle dorsiflexor muscles. It prevents the patient from effectively swinging the leg during walking, causing an abnormal gait characterized by hip hitching and circumduction and toe catch. Walking speed in people with drop foot is often significantly reduced and the risk of stumbling or falling is high. The conventional treatment for drop foot is an ankle-foot orthosis (AFO). While AFOs are appropriate for many patients, in certain patient groups AFOs have significant limitations (e.g. in patients with strong spasticity, suffering from pronounced inversion, suffering from volume changes in the lower extremity, etc). An alternative way of treating drop foot is by means of functional electrical stimulation. Clinical studies evaluating the effectiveness of drop foot stimulation suggest that it provides many benefits to patients, such as an improved confidence in walking, increased walking speed and endurance, less effort during walking and reduced spasticity. Implantable systems such as ActiGait are considered therapeutic alternatives specifically for those patients for whom conventional treatments have failed. ActiGait system consists of an external module (antenna and control module), a foot switch transmitting to the external module and an implanted assembly (receiver, pulse train generator, electrodes). The objective of this study is to obtain additional evidence on safety of ActiGait implantation procedure and on its efficacy. The study will enrol 5 subjects that will be implanted and followed for 12 weeks. Efficacy outcomes will be assessed at the baseline and during two follow-up visits (week 6 and 12). Subjects will be asked to walk with and without their preferred walking at the baseline and with and without stimulation at follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* have a single sided hemiparesis persisting for more than 6 months due to a cerebro-vascular accident (CVA).
* be fully grown-up.
* have the ability to walk 20 meters in less than 2 minutes with or without walking aid but without the help of another person.
* have a reduced speed of walking.
* have the ability to stand upright with both heels touching the floor while hip and knee are in neutral position.
* have a passive range of movement of the affected ankle joint of at least 30 degrees.
* have a positive response to surface electrical stimulation of the peroneal nerve - i.e. muscle contraction which results in dorsiflexion of the ankle and improved gait.
* male or female older than 18 years of age.
* have signed written Informed consent to participate in the study.
* is willing and able to follow all study procedures including attendance at clinics for scheduled study visits.

Exclusion Criteria:

* peripheral nerve damage of the affected leg.
* severe or uncontrolled diabetes with peripheral nerve involvement.
* poor skin condition on the affected leg.
* a thickness of subcutaneous fat exceeding 3.5 cm in the region of the implant.
* inability to walk 100 meters without stopping prior to CVA (with or without a walking aid, but without the help of another person).
* poorly controlled epilepsy.
* need of Ankle Foot Orthosis (AOF) to maintain ankle stability.
* concomitant medical and psychological conditions which would limit the success of the ActiGait® system such as: active degenerative diseases of the back and lower limbs, visuo-spatial neglect, or drug abuse, personality disorders or poor cognitive function.
* concomitant medical and psychological conditions which would compromise the safety of the patient in connection with the implantation and use of the ActiGait system, such as: severe cardiac disease, uncontrolled hypertension or history of malignancy within the preceding five years.
* other active implanted devices such as demand pacemakers or implanted defibrillators, as mutual electromagnetic interference may distort the efficacy of both systems and expose the patient to dangerous situations.
* history of falls greater than once a week.
* pregnancy and lactation. Women of childbearing potential must maintain effective contraception during the study period, as judged by the investigator.
* previous participation in this study
* participation in an investigational drug trial within 4 weeks prior to enrolment.
* requirement of an interpreter
* use of external FES system to assist walking four weeks prior to enrolment
* MRI of the affected thigh that is inconsistent with safe implantation of the ActiGait
* history of falls greater than once a week.
* pregnancy and lactation. Women of childbearing potential must maintain effective contraception during the study period, as judged by the investigator.
* previous participation in this study.
* participation in an investigational drug trial within 4 weeks prior to enrolment.
* requirement of an interpreter.
* anatomic situation of the common peroneal nerve identified by pre-surgical MRI that could compromise the success of ActiGait).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Liebetanz, MD, Principal Investigator — Medical University Georg-August-University Goettingen, Germany; Veit Rhode, MD, Principal Investigator — Medical University Georg-August-University Goettingen, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- ActiGait - Implantable Drop Foot Stimulator: Subjects came with conventional walking aid and then received ActiGait implant
Period: Overall Study
Arm/Group | ActiGait - Implantable Drop Foot Stimulator
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ActiGait - Implantable Drop Foot Stimulator
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Number; unit: participants]
  Germany | 5

OUTCOME MEASURES:

1. Primary Outcome: Distance Walked in 6 Minutes
Description: The test assesses distance walked over 6 minutes as a sub-maximal test of aerobic capacity (endurance). At baseline this test was done with subject's conventional walking aid. At 6 and 12 weeks post-implantation this was done with and without stimulation.
Time Frame: Baseline, 6 and 12 weeks post-implantation
Measure: Mean (Standard Deviation); unit: m
Arm/Group | ActiGait - Implantable Drop Foot Stimulator
Number analyzed (Participants) | 5
m
  Baseline | 211 (36.78)
  6 weeks post-implantation stimulation off | 211 (37.48)
  6 weeks post-implantation stimulation on | 260 (31.5)
  12 weeks post-implantation stimulation off | 214 (33.46)
  12 weeks post-implantation stimulation on | 248 (29.56)

2. Secondary Outcome: Walking Speed During 10 Meter Gait Test
Description: The test assesses walking speed in meters per second over a short duration. At baseline this test was done with subject's conventional walking aid. At 6 and 12 weeks post-implantation this was done with and without stimulation.
Time Frame: Baseline, 6 and 12 weeks post-implantation
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | ActiGait - Implantable Drop Foot Stimulator
Number analyzed (Participants) | 5
m/s
  Baseline | 0.62 (0.07)
  6 weeks post-implantation stimulation off | 0.55 (0.065)
  6 weeks post-implantation stimulation on | 0.77 (0.077)
  12 weeks post-implantation stimulation off | 0.55 (0.071)
  12 weeks post-implantation stimulation on | 0.77 (0.064)

3. Secondary Outcome: Canadian Occupational Performance Measure (COPM) Score
Description: A semi-structured interview is conducted in order to identify subject's limitations with daily occupations of importance in categories self-care, productivtiy or leisure. The subject is then asked to rate the imporance of each of the occupations using a 10-point rating scale. Afterwards the subject chooses up to 5 of the most important occupations (problems) (basis for identifying intervention goals). The subject is asked to use a 10 point scale to rate level of performance and satisfaction with performance for each of the five identified problems. Average COPM performance score and satisfaction score are calculated. The scores range between 1 and 10, where 1 indicates poor performance and low satisfaction, respectively, while 10 indicates very good performance and high satisfaction.
Time Frame: Baseline,12 weeks post-implantation
Population: Two subjects were not available for the test.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ActiGait - Implantable Drop Foot Stimulator
Number analyzed (Participants) | 3
units on a scale
  Performance Baseline | 3.37 (1.27)
  Performance 12 weeks post-implantation | 3.80 (1.74)
  Satisfaction Baseline | 2.47 (0.46)
  Satisfaction 12 weeks post-implantation | 2.70 (0.70)

4. Secondary Outcome: Four Square Step Test (FSST)
Description: It is a test of dynamic balance that clinically assesses the person's ability to step over objects forward, sideways, and backwards. The patient's time to perform the test is measured which shorter time representing better performance. At baseline this test was done with subject's conventional walking aid. At 12 weeks post-implantation it was done with and without stimulation.
Time Frame: Baseline, week 12 post-implantation
Measure: Mean (Standard Deviation); unit: s
Arm/Group | ActiGait - Implantable Drop Foot Stimulator
Number analyzed (Participants) | 5
s
  Baseline | 38.09 (27.41)
  12 weeks post-implantation stimulation off | 44.44 (39.51)
  12 weeks post-implantation stimulation on | 21.49 (5.54)

5. Secondary Outcome: Nerve Conduction Velocity of the Peroneal Nerve
Description: Measured: Nervus peroneus communis (CPN) and Nervus peroneus superficialis (SPN)
Time Frame: Baseline, week 12 post-implantation
Population: Two subjects were unavailable for the test.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | ActiGait - Implantable Drop Foot Stimulator
Number analyzed (Participants) | 3
m/s
  Baseline CPN | 48.33 (4.73)
  Baseline SPN | 43 (1)
  12 weeks post-implantation CPM | 50 (4.36)
  12 weeks post-implantation SPN | 42.67 (6.66)

6. Secondary Outcome: Change in MRI of Affected Leg and Implant Post-implantation
Description: MRI will be conducted to evaluate the impact of the implant on the common peroneal nerve (e.g. positioning of the nerve cuff along the nerve, path of the lead wire and the common peroneal nerve, estimation of the cross-sectional area of the common peroneal nerve compared to the pre-operative MRI recording, etc.).
  The outcome will be quantified by surgeon's judgement whether the final implant position is consistent with safe application of the ActiGait® implant as described in the manufacturer's surgical manual. Number of safe and successful implantations will be counted.
Time Frame: Week 2 post-implantation
Measure: Number; unit: number of safe implantations
Arm/Group | ActiGait
Number analyzed (Participants) | 5
number of safe implantations | 5

ADVERSE EVENTS:
Arm/Group | ActiGait - Implantable Drop Foot Stimulator
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ActiGait - Implantable Drop Foot Stimulator (N=5)
Haematoma around implantation site and bleeding after stitches removal, requiring additional surgery (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ActiGait - Implantable Drop Foot Stimulator (N=5)
Post-surgical lymphoedema around proximal incision (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No